CLINICAL TRIAL: NCT04848454
Title: Neoadjuvant Camrelizumab Combined to Vinorelbine and Cisplatin as Second Regimen to Non-optimal Response to Taxanes and Anthracyclines on Patients With Early Stage HER2-negative Breast Cancer: A Single Arm Phase 2 Trial
Brief Title: Efficacy and Safety of Combinition of Camrelizumab in Second-line Neoadjuvant Chemotherapy and Adjuvant Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, XU Ling, Chief Physician of Breast Disease Center, Associate Professor, M.D., Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-BB-BC-II-007
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: HER2-negative Breast Cancer; Neoadjuvant Therapy; Pathological Complete Response; Immunotherapy; Vinorelbine; Cisplatin
MeSH Terms: interventions — camrelizumab; Vinorelbine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Drug:
  Vinorelbine i.v. 25 mg/m2, d1, d8 or p.o. 60-80 mg/m2 d1, d8; q3w; for 6 cycles.
  Cisplatin i.v. 75 mg/m2，d1, d2; q3w; for 6 cycles. Camrelizumab i.v. 200mg, q3w; for 17cycles (1 year).
  Interventions: Drug: Camrelizumab with vinorelbine and cisplatin

INTERVENTIONS:
Drug: Camrelizumab with vinorelbine and cisplatin — Camrelizumab: 200mg iv., every 3 weeks(one cycle), for 1 year(17cycles in total); Vinorelbine: 25mg/m2 day 1, 8 iv. or 60-80 mg/m2 or. day1, 8, every 3 weeks(one cycle), for 6 cycles; Cisplatin: 75mg/m2 (divided into 2 days), every 3 weeks(onr cycle), for 6 cycles.

SUMMARY:
The achievement of pathological complete response (pCR) after neoadjuvant chemotherapy (NACT) is associated with improved outcome across all breast cancer (BC) subtypes. Anthracycline and taxanes based chemotherapy is usually the first choice of NACT for human epidermal growth factor receptor 2 (HER2) negative breast cancer, but there is no ideal second-line therapy for those with unsatisfactory effect after first-line NACT. Vinorelbine combined with cisplatin may be a choice for patients after failure or progression with anthracycline and/or taxanes. Immunotherapy has achieved good efficacy in many malignant tumors. Chemotherapy may have a certain immune activation effect, thus combination of immunotherapy and chemotherapy has significant clinical value in neoadjuvant and adjuvant treatment of breast cancer.

So we designed this one center single arm phase 2 clinical trial to test the efficacy and safety of camrelizumab (PD-1 inhibitor) combined with vinorelbine and cisplatin as a second-line therapy for HER2 negative breast cancer patients who did not achieve significant effect after 2 cycle treatments of anthracycline plus taxanes NACT.

The target population of our study are early-stage HER2 negative breast cancer patients with indications of NACT who did not receive partial response after 2 cycle of standard anthracycline and taxanes treaments according to RECIST 1.1 criteria. The enrolled patients will receive 6 cycles of camrelizumab combined with vinorelbine and cisplatin as second-line neoadjuvant therapy. Then they need to undergo surgery. The subjects have to continue camrelizumab until it is totally used for 1 year (about 17 cycles in all). The patients will routinely receive conventional adjuvant therapy and enter the long-term follow-up to get their survival infoumation.

DETAILED DESCRIPTION:
It has been proved that the achievement of pathological complete response (pCR) after neoadjuvant chemotherapy (NACT) is associated with improved outcome across all breast cancer (BC) subtypes. At present, anthracycline and taxanes based chemotherapy is usually the first choice of neoadjuvant therapy for human epidermal growth factor receptor 2 (HER2) negative breast cancer, and the response rate can be more than 2/3. However, there are still some patients not getting satisfactory outcome using this regimen, for whom there is no unified ideal second-line neoadjuvant therapy to choose. Studies on metastatic BC have shown that vinorelbine combined with cisplatin has good efficacy and safety in the treatment of patients after failure or progression with anthracycline and/or taxanes. In other studies, patients with poor response to anthracycline and taxanes based NACT changed to NACT containing vinorelbine could obtain improved long-term survival. These results suggest that adjusting the neoadjuvant therapy according to the efficacy may bring more benefits to patients and vinorelbine combined with cisplatin is one of the second-line options for HER2 negative breast cancer who has been treated by the anthracycline and taxanes based NACT but not getting good efficacy.

Immunotherapy has achieved good efficacy in many malignant tumors. The US Food and Drug Administration (FDA) has approved the indications for the use of pembrolizumab ( an anti-PD-1 antibody) and atezolizumab (an anti -PD-L1 antibody) in patients with unresectable locally advanced or metastatic triple negative breast cancer. In neoadjuvant therapy, many studies have shown that the increase of pCR rate after NACT combined with immunotherapy, and the clinical benefit is obvious in the early stage. This was hypothesized that chemotherapy including anthracyclines or other drugs may have a certain immune activation effect, thus combination of immunotherapy and chemotherapy has significant clinical value in neoadjuvant and adjuvant treatment of breast cancer.

Based on the above background, we propose the hypothesis that camrelizumab combined with vinorelbine and cisplatin can be recommended for HER2 negative breast cancer patients who did not achieve significant efficacy after 2 cycle treatments of anthracycline plus taxanes as first-line neoadjuvant therapy. In order to confirm this hypothesis, we designed the following one centre single arm phase 2 clinical trial.

We defined the target population of our study as those early-stage HER2 negative breast cancer (triple negative breast cancer and HER2 negative hormone receptor positive breast cancer) patients with indications of NACT who did not receive partial response after 2 cycle of standard anthracycline and taxanes treaments according to RECIST 1.1 criteria. We expect to recruit 30 subjects. The enrolled patients will receive 6 cycles of neoadjuvant therapy of camrelizumab combined with vinorelbine and cisplatin (NP) as second-line neoadjuvant therapy. After the patients complete the neoadjuvant therapy or stop treatment due to disease progression, intolerance of adverse reactions or other conditions that the researchers thought they could not continue to benefit from the treatment, they need to undergo surgery in 4 weeks. The subjects have to continue camrelizumab every 3 weeks like during the preoperative phase until it is totally used for 1 year (about 17 cycles in all). In addition, the patients will routinely receive conventional treatment, endocrine therapy and other adjuvant therapy. Our primary objection is to evaluate the efficacy of second-line neoadjuvant therapy with camrelizumab combined with NP; and the secondary objection is to verify this regimen's security. The efficacy of camrelizumab and NP neoadjuvant therapy will be evaluated according to the assessment during treatment, postoperative pathological results and follow-up results. We will record the clinical response, pCR, progression-free survival and overall survival etc. Safety information will be collected continuously at the beginning of study treatment until the completion of follow-up after study treatment. Besides, we will do some exploratory research using the histological or blood samples of the subjects about biomarkers (like tumor infiltrating lymphocytes, expression of PD-L1 etc.) that may be used for clinical prediction, selection of suitable population and other situations.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to join the trial and the follow-up; provide written informed consent.
* Be a male or female subject at the age when signing the informed consent of 18-70 years old.
* Have invasive breast cancer confirmed by histopathology, HER2 negative and suitable for neoadjuvant therapy (clinical stage is II or III).
* With at least one mearsurable lesions according to RECIST 1.1 criteria.
* No significant early response to first-line neoadjuvant therapy with anthracyclines and taxanes. Definition: first-line neoadjuvant regimen mainly refers to regimen: intravenous infusion of epirubicin 75mg/m2 day 1 or pirarubicin 60mg/m2 day 1 or liposome doxorubicin 25-35mg/m2 day 1, docetaxel 75mg/m2 day 2 or paclitaxel 135-175mg/m2 day 2 or albumin paclitaxel 200-260mg/m2 day 2, once every 3 weeks. After 2 cycles of treatment, the tumor size did not reach partial response (defined as the sum of the target lesion diameter decreased by at least 30% compared with the baseline), and second-line neoadjuvant therapy was considered.
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have an estimated life expectancy more than 6 months.
* Have adequate organ function, including: ① Bone marrow reserve (not using any blood components or cell growth factors within 14 days): WBC≥4.0×10^9/L, NEUT ≥ 1.5×10^9/L, PLT≥100×10^9/L, HGB≥100g/L; ② Hepatic function: ALT, AST≤2.5 ULN, total bilirubin≤ 1.5ULN; ③Renal function: Serum Creatinine≤1.5 ULN or creatinine clearance rate ≥50ml/min (Cockcroft Gault formula); ④ Has normal cardiac function as evidenced by an left ventricular ejection fraction (LVEF) ≥50% by echocardiogram. No obvious abnormal case in electrocardiogram. ⑤Female subjects of child-bearing age must carry out serum pregnancy test within 3 days before starting the study treatment, and the result must be negative, and they have to use a highly effective contraceptive measure (such as intrauterine device, contraceptive or condom) approved by medicine during the study period and within 3 months after the last administration of the study drug; for male subjects with female partners of child-bearing age, they should agree to use the contraceptive measure during the study period and within 3 months after the last study drug treatment .

Exclusion Criteria:

* Has any evidence of metastatic disease.
* Has received chemotherapy, targeted therapy, endocrine therapy or local radiotherapy in the past.
* Previously received anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell costimulation or checkpoint pathway).
* A clear history of allergy may lead to potential allergy or intolerance to the study drug and its similar biological agents.
* Participated in clinical trials of other anti-tumor drugs within 4 weeks before the first administration; or received live attenuated vaccine within 4 weeks before the first administration or planned during the study period.
* Had other malignant tumors occurred within 5 years (except for completely treated squamous cell carcinoma of skin or controlled basal cell carcinoma of skin).
* Immunosuppressive drugs were used within 14 days before the first use of camrelizumab, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e. not more than 10 mg/day of prednisolone or other corticosteroids of the same pharmacophysiological dose).
* Active autoimmune disease or history of autoimmune disease: including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma in childhood had complete remission and did not need any intervention in adulthood could be included; asthma that needs bronchodilator for medical intervention cannot be included.
* Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥450ms in male and ≥470ms in female); NYHA grade III-IV heart failure, or left ventricular ejection fraction (LVEF) < 50% by echocardiography; myocardial infarction within 6 months; NYHA grade I-II, uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease; ECG showed acute ischemia or active abnormality of conduction system.
* Severe infection occurred within 4 weeks before the first administration (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs) or fever of unknown origin > 38.5 ℃ occurred during the screening period or before the first administration.
* History of psychotropic substance abuse and can not give up or have mental disorders.
* Major surgery performed within 4 weeks before the first administration; with open wound or fracture;
* The adverse reactions related to anti-tumor therapy (except alopecia) did not return to nci-ctcae ≤ 1 after first-line neoadjuvant therapy.
* Other circumstances judged by the researchers not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 1 month after the definitive surgery (if the patient does receive the surgery, usually 3-4 weeks after the last cycle of neoajuvant therapy)
  The rate of pCR use the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) as assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 month after the last cycle of neoadjuvant therapy
  The rate of patients with complete remission (CR) or partial response (PR) evaluated by RECIST 1.1 criteria by site radiology review before operation.
Event-free survival (EFS) rate | 5 years
  The rate of patients in all assessable subjects without any of the following events: progression of disease that precludes surgery, local or distant recurrence (surgical complete resection of local lesion) , second primary malignancy (breast or other cancers) or death due to any cause.
Breast-conserving surgery rate | During the definitive surgery
  The rate of assessable patients undergoing breast-conserving surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China